CLINICAL TRIAL: NCT00744328
Title: Postpartum Depression: Transdermal Estradiol Versus Sertraline
Acronym: E2SERT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment Issues
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Katherine Wisner, Norman and Helen Asher Professor of Psychiatry and Behavioral Sciences and Obstetrics and Gynecology; Director, Asher Center for the Study and Treatment of Depressive Disorders, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH057102 (NIH)
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2018-08

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression; estradiol; Postpartum major depressive disorder
MeSH Terms: conditions — Depression, Postpartum | interventions — Estradiol; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transdermal Estradiol (Experimental): Women wear a skin patch that is changed weekly and take opaque capsules by mouth daily. The capsules for women in this arm do not contain any active ingredients. The skin patch contains transdermal estradiol ranging in dose from 50 to 200 mcg/day
  Interventions: Drug: Transdermal Estradiol; Other: Placebo
- Sertraline (Active Comparator): Women wear a skin patch that is changed weekly and take opaque capsules by mouth daily. The skin patch contains no active ingredients, though packaging is designed to match active patches. The capsules contain sertraline ranging in dose from 25 to 200mg/day
  Interventions: Drug: Sertraline; Other: Placebo
- Placebo (Placebo Comparator): Women wear a skin patch that is changed weekly and take opaque capsules by mouth daily. The capsules for women in this arm do not contain any active ingredients. The skin patch contains no active ingredients, though packaging is designed to match active patches.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Transdermal Estradiol — Estradiol patch ranging in dose from 50 to 200 mcg/day
  Other Names: Vivelle dot; Climara
  Arms: Transdermal Estradiol
Drug: Sertraline — Sertraline dose will range from 50 - 200 mg/day
  Other Names: Zoloft
  Arms: Sertraline
Other: Placebo — Placebo patches and pills that are identical to transdermal estradiol and oral sertraline, respectively, will be used.

SUMMARY:
The purpose of this study is to determine whether estrogen patches are effective for the treatment of postpartum major depression, as compared to sertraline (Zoloft) and placebo.

DETAILED DESCRIPTION:
This study aims to advance our therapeutic armamentarium by evaluating the efficacy of estradiol (E2) therapy for Postpartum Major Depression (PPMD), which has received minimal research attention in America. The design of the proposed study is an 8 week randomized double-blind clinical trial of SERT vs. E2 vs. Placebo. Responders enter a continuation phase with the blind intact through 6.5 months postpartum. The primary aims of this investigation are to: 1) Test the efficacy of E2 compared to placebo for the treatment of PPMD. Sertraline will be included as an active comparator. We have powered the study to test for differences among the three groups and also test for differences between the E2 and placebo group. We will test the hypothesis that E2 will be significantly more effective than placebo and that SERT will be significantly more effective than placebo. 2) Evaluate developmental outcomes in infants exposed to the disorder, PPMD, and the medications (SERT, exogenous E2 or Placebo) which may be transmitted to the infants through breastfeeding. All infants in this study will have exposure to mothers with depression. We will assess maternal depression, mother-infant serum SERT and E2 levels and relate them to mother-infant interactional quality and infant developmental outcomes on the Bayley Scales of Infant Development. These data will enhance the sophistication of risk-benefit analyses for pharmacotherapy during lactation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45 years
* Had a baby within the last 3 months
* Experiencing depression or lasting sadness

Exclusion Criteria:

* Current use of other therapies for depression, such as antidepressants, psychotherapy, bright light therapy, and herbal remedies such as Hypericum St. John's Wort
* DSM-IV diagnoses of bipolar 1 or 2 disorder or any psychotic episode; substance abuse within last 6 months
* Previous adverse reaction to sertraline or provera
* No pediatric care: No pediatrician with whom to coordinate breastfeeding and infant care
* Use of medications for medical disorders, except for treatment of hypothyroidism or inhalers for asthma or progestin-only contraceptives
* Heavy smoking (>10 cigarettes per day) or intent to resume heavy smoking (unless willing to cut down)
* personal history of thromboembolic event, hypercoagulability, or first degree relatives with thromboembolic events.
* Current or past personal history of breast, uterine, or ovarian cancer.
* BRCA-positive mother
* Arterial vascular disease and/or heart disease: increased risk of stroke.
* Liver disease: increased risk of biliary stones, cholestatic jaundice and benign hepatic lesions with E2 treatment.
* Diabetes
* Pregnancy
* Infants born <32 weeks of gestation
* Imminent suicidality and/or homicidality: in need of higher level of care than is provided in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2008-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Wisner, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine; Asher Center for the Study and Treatment of Depressive Disorders, Chicago, Illinois, United States

REFERENCES:
- [Derived] Pulido CM, Walson IS, Yang A, Stika CS, Sit DK, Wisner KL. Differentiating Depressive Symptoms From Side Effects in Individuals With Major Depressive Disorder With Postpartum Onset. J Clin Psychopharmacol. 2025 Mar-Apr 01;45(2):106-110. doi: 10.1097/JCP.0000000000001928. Epub 2024 Dec 4. PMID 39626074
- [Derived] Prairie BA, Wisniewski SR, Luther JF, Sit D, Wisner KL. Postpartum lipid levels in women with major depression. J Womens Health (Larchmt). 2012 May;21(5):534-8. doi: 10.1089/jwh.2011.3256. Epub 2012 Jan 27. PMID 22283499
- See also: Northwestern Psychiatry Homepage — http://psychiatry.northwestern.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol: Administered via skin patch ranging in dose from 50 to 200 mcg/day
  Transdermal Estradiol: Estradiol patch ranging in dose from 50 to 200 mcg/day
- Sertraline: Administered via capsules taken orally ranging in dose from 25 to 200mg/day
  Sertraline: Sertraline dose will range from 50 - 200 mg/day
Period: Overall Study
Arm/Group | Estradiol | Sertraline | Placebo
Started | 26 | 30 | 29
Completed | 19 | 22 | 21
Not Completed | 7 | 8 | 8
Not completed — Lost to Follow-up | 2 | 5 | 3
Not completed — Withdrawal by Subject | 5 | 3 | 4
Not completed — Found ineligible after randomization | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol | Sertraline | Placebo | Total
Number analyzed (Participants) | 26 | 30 | 29 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.98) | 26.2 (5.89) | 27.4 (5.48) | 26.6 (5.74)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 30 | 29 | 85
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 29 | 85
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 10 | 9 | 4 | 23
  White | 14 | 19 | 21 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 26 | 30 | 29 | 85
SIGHADS29 [Mean (Standard Deviation); unit: Scores on a scale] — Depression was assessed with the Structured Interview Guide for the Hamilton Depression Rating Scale - Atypical Depression Symptoms Version (SIGH-ADS29). The scale incorporates the 17 and 21-item Hamilton Rating Scales for Depression (HRSD) as well as 8 atypical symptoms of depression. Scores range from 0 to 90, where a higher score corresponds to a higher level of depressive symptomatology. A minimum SIGH-ADS29 score of 18 was required for enrollment.
  Scores on a scale | 23.3 (4.99) | 23.3 (3.67) | 25.1 (4.92) | 23.9 (4.56)

OUTCOME MEASURES:

1. Primary Outcome: To Test the Efficacy of Estradiol for the Treatment of Postpartum Depression - Percent Change in SIGH-ADS29
Description: Depression was assessed with the Structured Interview Guide for the Hamilton Depression Rating Scale - Atypical Depression Symptoms Version (SIGH-ADS29). The scale incorporates the 17 and 21-item Hamilton Rating Scales for Depression (HRSD) as well as 8 atypical symptoms of depression. Scores range from 0 to 90, where a higher score corresponds to a higher level of depressive symptomatology.
Time Frame: Week 8
Population: Analyses presented are Last Observation Carried Forward. For women who completed the 8 week trial the percent change was measured from baseline to week 8. For non-completers, the percent change was measured from baseline to last observation.
Measure: Mean (Standard Deviation); unit: percentage change in SIGH-ADS29 Score
Arm/Group | Estradiol | Sertraline | Placebo
Number analyzed (Participants) | 26 | 30 | 29
percentage change in SIGH-ADS29 Score | -38 (33.7) | -49 (24.1) | -48 (29.8)

2. Secondary Outcome: Infant Serum Concentrations of Estradiol in 3 Treatment Arms
Description: As expected due to being stopped and therefore underpowered
Time Frame: monthly
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol | Sertraline | Placebo
Number analyzed (Participants) | 6 | 6 | 7
pg/mL | 2.45 (3.80) | 2.1 (3.36) | 5.59 (7.79)

ADVERSE EVENTS:
Time Frame: Weekly during the 8-week acute phase
Description: If a patient develops a symptom score on the Mania Rating Scale of >10, she will receive an immediate consultation for a revised treatment regimen by non-blind medical monitor to keep primary study staff blind to pill/patch content. Occurrence of hypomania/mania will signal termination from the trial.
Arm/Group | Estradiol | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/26 | 4/30 | 1/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol (N=26) | Sertraline (N=30) | Placebo (N=29)
Treatment Emergent Manic Symptoms (Psychiatric disorders) | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No